CLINICAL TRIAL: NCT04531423
Title: PKC as Serum Biomarkers for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: smhcgxy
Record Dates: First submitted 2020-08-16; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; golimumab

STUDY DESIGN:
Intervention Model Description: The investigators adopted randomized design to test placebo-controlled antidepressant augmentation.Participants were randomized (1:1) into one of the following 2 groups: "SSRI +golimumab"," or "SSRI +placebo".
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSRI + golimumab (Experimental): Participants will be administered with SSRI+golimumab . Golimumab will be administered at the dose of 50mg every month during the acute phase.
  Interventions: Drug: SSRI + golimumab
- SSRI +placebo (Active Comparator): Participants will be administered with SSRI+placebo
  Interventions: Other: SSRI + placebo

INTERVENTIONS:
Drug: SSRI + golimumab — Golimumab will be administered at the dose of 50mg every month during the acute phase.
  Arms: SSRI + golimumab
Other: SSRI + placebo — placebo
  Arms: SSRI +placebo

SUMMARY:
Inflammation that is mediated by microglia activation plays an important role in the pathogenesis of depression. Microglia activation can lead to an increase in the levels of proinflammatory cytokines, including TNF-α, which leads to neuronal apoptosis in the specific neural circuits of some brain regions, abnormal cognition, and treatment-resistant depression (TRD). Protein kinase C (PKC) is a key regulator of the microglia activation process. The investigators assume that the abnormality in PKC might be the serum biomarkers of depression.

DETAILED DESCRIPTION:
PKC activation might reduce M1 microglia activation and the release of proinflammatory cytokines such as TNF-α, finally alleviating depressive symptoms in TRD.

Primary objective: This study was designed to address the role of PKC-mediated microglial activation in the clinical outcome of first episode depression.

Secondary objective: To illustrate the impact of PKC-mediated microglial activation on impaired cognition, social function and neuronal plasticity.

The investigators adopted randomized design to test placebo-controlled antidepressant augmentation. Patients were randomized (1:1) into one of the following 2groups: "SSRI +golimumab"," or "SSRI +placebo". The total study duration is 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);

  * Insufficient response (response rate <50%) to two antidepressants with different mechanisms when given for at least 6 weeks at an adequate dose (e.g., clomipramine ≥150 mg/d, fluoxetine≥20 mg/d) during the current episode;

    * A 17-item Hamilton Depression Rating Scale (HAMD-17) score ≥ 17 no more than 7 days prior to randomization. Cognitive factors (including a sense of guilt, suicidal thoughts, agitation, depersonalization, the disintegration of reality, paranoid symptoms, and obsessive and compulsive symptoms) score ≥6; ④ Between 18 and 65 years of age;

      ⑤ Education: finished junior middle school;

      ⑥ Ethnicity: Han Chinese;
      * Adequate audio and visual levels to complete the necessary checks; ⑧ Compliance with treatment in the clinical trial.

Exclusion Criteria:

* Severe liver and kidney diseases, active endocrine diseases or clinical symptoms. Severe cardiovascular disease, respiratory system disease, hematologic diseases and cancer.

  * Serious suicide attempts.

    * Pregnancy or lactation.

      * Modified electroconvulsive therapy (MECT) therapy in the past 1 month. ⑤ Known current psychosis as determined by the DSM-5 or a history of a non-mood psychotic disorder.

        * Participation in another clinical trial concurrently or no more than 1 month prior to randomization.

          * Previously had a severe allergic reaction or immune system disease; ⑧ Using an anti-inflammatory drug or immunosuppressive agent; ⑨ HAMD-17 item 3 (suicide) score: ≥3

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 12 weeks
  The primary outcome is defined as changes in HAMD-17 between baseline and 12weeks scored 7 or lower on the Hamilton's Depression Scale with 17 items

IPD SHARING:
Plan to Share IPD: No